CLINICAL TRIAL: NCT07334964
Title: Ultrasound-Guided Carpal Tunnel Infiltration: Comparison Between the Manual Method and a Robot-Assisted Method - A Pilot, Comparative, Randomized Study
Brief Title: Ultrasound-Guided Carpal Tunnel Infiltration: Comparison Between the Manual Method and a Robot-Assisted Method
Acronym: ICCERO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUO-2025-06
Record Dates: First submitted 2025-12-22; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; robot-assited-ultrasonography; carpal tunnel injection
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: There are 2 arms with an equal number of patient randomized in a parallel way.
Who Masked: Participant
Masking Description: blinding during injection: a vertical drape blocking the view between the operator and the participant; the robot activated in both groups (noise), noise-reduction system for the patient (noise-canceling headset on the participant's ears, use of earphones, etc.), nurse present in both groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual (Arm A) (Active Comparator): Ultrasound-guided carpal tunnel injection using the conventional method:
  An ultrasound-guided carpal tunnel injection is performed using manual guidance. The operator first identifies the median nerve using an ultrasound probe. The operator then applies aseptic conditions. Subsequently, the operator holds the ultrasound probe in one hand and the medication in the other, and performs the injection while referring to the ultrasound image to ensure accurate needle placement.
  Interventions: Procedure: Carpal tunnel injection
- Robot-Assisted (Arm B) (Experimental): Ultrasound-guided carpal tunnel injection assisted by a robotic arm:
  The operator first identifies the median nerve using an ultrasound probe tied back to the robotic arm. The operator then places both themselves and the probe attached robotic arm under aseptic conditions. The robotic arm is subsequently positioned to obtain the desired ultrasound imaging plane. The operator then has both hands free to perform the injection, referring to the ultrasound image to ensure accurate needle placement.
  Interventions: Procedure: Carpal tunnel injection

INTERVENTIONS:
Procedure: Carpal tunnel injection — Ultrasound localization will be performed by the physician. He will then perform the injection under ultrasound guidance. In Group A, maintenance of the ultrasound probe during the injection will be performed by the physician assisted by a nurse. In Group B, maintenance of the ultrasound probe during the injection will be performed by the robotic arm.
  All other aspects of the procedure will be carried out according to usual standards (localization, aseptic technique, injection, etc…). The procedure will be timed from the initial positioning (first contact of the ultrasound probe with the wrist) to the end of the injection (needle withdrawal).
  Maintenance of participant blinding during the injection: a drape will be placed between the physician and the participant; the robot will be activated in both groups, the participant will wear anti noise headphones, and a nurse will be present in both groups.

SUMMARY:
This study aims to assess the feasibility, safety, and accuracy of a robotic arm-assisted carpal tunnel injection in comparison with the conventional ultrasound-guided method, prior to conducting a larger-scale study.

The use of a robotic arm to maintain the ultrasound probe in position could provide valuable assistance to the physician. The procedure would no longer require the involvement of a third person in addition to the physician. To date, no study has compared these two approaches.

DETAILED DESCRIPTION:
This study will be offered to patients suffering from carpal tunnel syndrome who are followed for this condition in a rheumatology setting. The carpal tunnel injection, as well as identification of the injection site using an ultrasound probe, will be performed by the practitioner according to standard clinical practice.

Maintaining the ultrasound probe during the injection will constitute the research-specific procedure (standard practice in Group A versus a research-specific procedure with probe holding by the robotic arm in Group B). Follow-up visits (at Day 7, Day 28 and 3 months after carpal tunnel injection) conducted via phone call, teleconsultation or consultation will also be research-specific procedures, as will completion of the pain VAS (Visual Analogue Scale), the BQCT (Boston carpal tunnel syndrome questionnaire) self-administered questionnaire, and the participant satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years.
2. Clinical diagnosis of carpal tunnel syndrome.
3. Indication for corticosteroid injection as determined by investigator.
4. Moderate to severe carpal tunnel syndrome defined by a pain score on the Visual Analogue Scale (VAS) ≥ 4 (at baseline and on day 0).
5. Signed informed consent.

Exclusion Criteria:

1. Known allergy to corticosteroids or povidone-iodine (Betadine)
2. Probable or ongoing systemic or local infection
3. History of injection in the affected wrist within the last 6 months
4. Thenar eminence atrophy
5. Trauma requiring surgery or immobilization
6. History of carpal tunnel surgery
7. Protected person (under guardianship or curatorship)
8. Person under judicial protection
9. Person deprived of liberty
10. Person not affiliated with a social security scheme
11. Pregnant or breastfeeding woman
12. Person participating in a drug trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-11-25 (Estimated); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
Comparison of the variation of the VAS scale on the Ultrasound-Guided Carpal Tunnel Injection between the Manual Method and a Robot-Assisted Method | This outcome is measured on the day of the intervention (Day 0) after randomization and a month after the intervention (Day 28)
  VAS: Scale 1 to 10 with 1 is no pain at all and 10 is the worst pain that the participant can imagine.

SECONDARY OUTCOMES:
Pain VAS at D7 and 3 months | This outcome is measured on Day 0 (D0) after randomization, Day 7 (D7), Day 28 (D28), and Month 3 (M3)
  VAS: Scale 1 to 10 with 1 is no pain at all and 10 is the worst pain that the participant can imagine.
Compare the evolution of the BCTQ (Boston Carpal Tunnel Questionnaire, subscale SSS) score over time according to the method (Arm A versus Arm B) | This outcome is measured on Day 0 (D0) after randomization, Day 7 (D7), Day 28 (D28), and Month 3 (M3)
  Compare the evolution of the Symptom Severity Scale (SSS) score, subscale 1 of BCTQ score. This subscale, the minimum is 11 points (no symptoms) and the maximum is 55 points (maximum severity of symptoms).
Compare the evolution of the BCTQ (Boston Carpal Tunnel Questionnaire, subscale FSS) score over time according to the method (Arm A versus Arm B) | This outcome is measured on Day 0 (D0) after randomization, Day 7 (D7), Day 28 (D28), and Month 3 (M3)
  Compare the evolution of the Functional Status Scale (FSS) score, subscale 2 of BCTQ score. This subscale, the minimum is 8 points (no functional difficulty) and the maximum is 40 points (maximum functional difficulties).
Compare the duration of the procedure according to the method (Arm A versus Arm B) | This outcome is measured on Day 0 (D0) after randomization
  Procedure duration, in minutes, measured between initial positioning (first contact of the ultrasound probe with the wrist) and completion of the injection (needle withdrawal).
Assess the procedure related pain | This outcome is measured n Day 0 (D0) after randomization and Day 7 (D7),
  Procedure-related pain measured at D0 immediately after the procedure using a pain VAS; and occurrence of complications such as hematoma or inflammatory reaction, assessed at D7. For VAS scale, the minimum value is 0 (no pain) and the maximum value is 10 (worst pain imaginable)
Assess patient satisfaction ("appreciation") regarding the robotic arm | This outcome is measured on Day 0 (D0) after randomization an before the procedure (carpal tunnel injection)
  Patient satisfaction ("appreciation") questionnaire regarding the robotic-assisted procedure at D0 (before the procedure). The "questionnaire d'appréciation de la procédure robotisée" questionnaire is specific for this study.
Assess the acceptability of patients participating in the study | This outcomme i measured at the end of the study
  Number of patients screened (inclusion visit), number of patients who agreed to participate in the study.
Compare analgesic consumption related to carpal tunnel syndrome over time | This outcome is measured on Day 0 (D0) after randomization, Day 7 (D7), Day 28 (D28), and Month 3 (M3)
  Analgesic consumption (number/type/frequency), including step 1-3 analgesics, tricyclic antidepressants, and gabapentinoids, assessed at D0, D7, D28, and M3.

CONTACTS AND LOCATIONS:
Overall Officials: Camille LANGBOUR, Dr, Principal Investigator — CHU Orléans
Locations (1):
- CHU Orléans, Orléans, France

REFERENCES:
- [Background] Lam KHS, Wu YT, Reeves KD, Galluccio F, Allam AE, Peng PWH. Ultrasound-Guided Interventions for Carpal Tunnel Syndrome: A Systematic Review and Meta-Analyses. Diagnostics (Basel). 2023 Mar 16;13(6):1138. doi: 10.3390/diagnostics13061138. PMID 36980446
- [Background] Goswami RP, Sit H, Chatterjee M, Lahiri D, Sircar G, Ghosh P. High-resolution ultrasonography in carpal tunnel syndrome: role of ancillary criteria in diagnosis and response to steroid injection. Clin Rheumatol. 2021 Mar;40(3):1069-1076. doi: 10.1007/s10067-020-05228-8. Epub 2020 Jul 21. PMID 32696280
- [Background] Lee JY, Park Y, Park KD, Lee JK, Lim OK. Effectiveness of ultrasound-guided carpal tunnel injection using in-plane ulnar approach: a prospective, randomized, single-blinded study. Medicine (Baltimore). 2014 Dec;93(29):e350. doi: 10.1097/MD.0000000000000350. PMID 25546691
- [Background] Mehta SP, Weinstock-Zlotnick G, Akland KL, Hanna MM, Workman KJ. Using Carpal Tunnel Questionnaire in clinical practice: A systematic review of its measurement properties. J Hand Ther. 2020 Oct-Dec;33(4):493-506. doi: 10.1016/j.jht.2019.12.011. Epub 2020 Mar 7. PMID 32151499
- [Background] Leite JC, Jerosch-Herold C, Song F. A systematic review of the psychometric properties of the Boston Carpal Tunnel Questionnaire. BMC Musculoskelet Disord. 2006 Oct 20;7:78. doi: 10.1186/1471-2474-7-78. PMID 17054773
- [Background] Jiang A, Qian Y, Yan J, Zhang S, Zhu S. Corticosteroid injection for carpal tunnel syndrome: A meta-analysis comparing ultrasound guided approach with landmark approach. Pak J Med Sci. 2024 Mar-Apr;40(4):773-778. doi: 10.12669/pjms.40.4.8749. PMID 38545011
- [Background] Priester AM, Natarajan S, Culjat MO. Robotic ultrasound systems in medicine. IEEE Trans Ultrason Ferroelectr Freq Control. 2013 Mar;60(3):507-23. doi: 10.1109/TUFFC.2013.2593. PMID 23475917
- [Background] Scheibert A, Preuss M, Osburg J, Ernst F, Kleemann M, Horn M. Robotic Assisted Ultrasound-Guided Endovascular Stent Implantation in a Vascular Model. Int J Med Robot. 2024 Dec;20(6):e70005. doi: 10.1002/rcs.70005. PMID 39501897
- [Background] Eilers C, van Kemenade R, Busam B, Navab N. On the importance of patient acceptance for medical robotic imaging. Int J Comput Assist Radiol Surg. 2023 Jul;18(7):1261-1267. doi: 10.1007/s11548-023-02948-5. Epub 2023 May 29. PMID 37248427
- [Background] Peters-Veluthamaningal C, Winters JC, Groenier KH, Meyboom-de Jong B. Randomised controlled trial of local corticosteroid injections for carpal tunnel syndrome in general practice. BMC Fam Pract. 2010 Jul 29;11:54. doi: 10.1186/1471-2296-11-54. PMID 20670438